CLINICAL TRIAL: NCT06220487
Title: A Single-arm, Open-label Study of Olverembatinib, CD3/CD19 Bispecific T-cell Engager, and Chidamide in Patients With Newly Diagnosed Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia
Brief Title: A Single-arm, Open-label Study of Olverembatinib, CD3/CD19 Bispecific T-cell Engager, and Chidamide in Patients With Newly Diagnosed Ph+ALL
Acronym: ABC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2023-441
Record Dates: First submitted 2023-12-03; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Acute Lymphoblastic Leukemia; Philadelphia Chromosome; Philadelphia-Positive ALL; Adult ALL; IKZF1 Gene Mutation
Keywords: Olverembatinib; CD3/CD19 Bispecific T-cell Engager; Histone Deacetylase Inhibitor; Chidamide; Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia; Ph-positive
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Philadelphia Chromosome | interventions — Prednisone; olverembatinib; blinatumomab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ABC protocol (Experimental): Adult patients with Ph-positive ALL eligble for this study will begin treatment with ABC protocol, as (A) olverembAtinib, (B) Blinatumomab and (C) Chidamide after pre-treatment with glucocorticoid, including induction and consolidation therapy for one year, and subsequent maintenance therapy for three years.
  Interventions: Drug: Prednisone, Olverembatinib, Blinatumomab, Chidamide

INTERVENTIONS:
Drug: Prednisone, Olverembatinib, Blinatumomab, Chidamide — Phase One. Induction Consolidation, for 1 year. 1.1 Pretreatment ×1 cycle. Prednisone，1mg/kg/d, from day 1 to 14;
  1.2 Induction Therapy × 1 cycle. A: OlverembAtinib (at a dose of 40 mg Qod), from day 8 to 42. B: Blinatumomab (at a dose of 28 μg per day), from day 15 to 28. C: Chidamide (at a dose of 10 mg Qod), from day 9 to 41.
  1.3 Consolidation Block × 5 cycles. A: Olverembatinib (at a dose of 40 mg Qod) was administered from day 1 to 42. B: Blinatumomab (at a dose of 28 μg perday) was administered from day 1 to 14. C: Chidamide (at a dose of 10 mg Qod) was administered from day 14 to 41.
  Phase Two. Maintenance Therapy, for 3 years. 2.1 A: Olverembatinib (at a dose of 40 mg Qod) was administered from day 1 to 42.
  C: Chidamide (at a dose of 10 mg Qod) was administered from day 14 to 41.
  Phase Three. Follow-up, for 5 years.

SUMMARY:
ABC study is a phase 2, single-arm, open-label study of Olverembatinib, CD3/CD19 Bispecific T-cell Engager, and Chidamide in patients with newly diagnosed Philadelphia Chromosome-positive acute lymphoblastic leukemia (Ph+ALL). This study combined third generation TKI (Olverembatinib), histone deacetylase inhibitors (Chidamide) and CD3/CD19 bispecific T-cell engager (Blinatumomab) as first line regimen (ABC regimen) for Ph+ ALL. Investigatorsaim to explore the efficacy and safety of ABC regimen. The primary endpoint is the complete molecular remission （CMR） at 3 months, secondary endpoints are overall survival (OS), event-free survival (EFS), adverse event (AE), IKZF1del, IKZF1plus, IKZF1lpus/CD20 subgroup EFS/OS.

DETAILED DESCRIPTION:
Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ALL) is now a relatively favorable-risk leukemia with the development of potent BCR::ABL1 tyrosine kinase inhibitors (TKIs). Achievement of an early and deep complete molecular remission (CMR) is an important end point in Ph+ ALL and identifies patients who may not need allogeneic hematopoietic stem cell transplantation (allo-HSCT). The chemotherapy-free D-ALBA trial of dasatinib and blinatumomab was safe and effective in patients with newly diagnosed Ph-positive ALL and resulted in an estimated 3-year OS rate of 80% (NEJM 2020, 2022). To further improve the outcomes, the potent third-generation TKIs, ponatinib and olverembatinib (ASH 2023, abs 1504), were added to chemotherapy or immunotherapy, resulted in an overall CMR rate of 84%-90%, a 5-year survival rate of 73%, most patients did not undergo allo-HSCT.

Of note, IKZF1plus subgroup still stands for high-risk for Ph+ALL and exhibit poor outcome even in TKI plus blinatumomab, which indicate IKZF1del confers resistance to immunotherapy. our previous study found that HDACi tucidinostat/chidamide could restore the expression and functionality of IKZF1 in IKZF1del samples, including increased expression of CD19 and reduced focal adhesion (Blood (2021) 138 (Supplement 1): 514.).

ABC study is a phase 2, single-arm, open-label study of Olverembatinib, CD3/CD19 Bispecific T-cell Engager, and Chidamide in patients with newly diagnosed Philadelphia Chromosome-positive acute lymphoblastic leukemia (Ph+ALL). This study combined third generation TKI (Olverembatinib), histone deacetylase inhibitors (Chidamide) and CD3/CD19 bispecific T-cell engager (Blinatumomab) as first line regimen (ABC regimen) for Ph+ ALL. Investigators aim to explore the efficacy and safety of ABC regimen. The primary endpoint is the complete molecular remission （CMR） at 3 months, secondary endpoints are overall survival (OS), event-free survival (EFS), adverse event (AE), IKZF1del, IKZF1plus, IKZF1lpus/CD20 subgroup EFS/OS.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Newly diagnosed adult B-precursor Ph+ ALL;
3. Age greater or equal to 18 years;
4. ECOG Performance Status 0-1;
5. Ineligible for allo-HSCT.
6. Renal and hepatic function as defined below:

   AST (GOT), ALT (GPT), and AP <2 x upper limit of normal (ULN). Creatinine clearance equal or greater than 50 mL/min.
7. Pancreatic function as defined below:

   Serum amylase less or equal to 1.5 x ULN Serum lipase less or equal to1.5 x ULN
8. Normal cardiac function;
9. Negative HIV test, negative HBV DNA and HCV RNA;
10. Negative pregnancy test in women of childbearing potential.

Exclusion Criteria:

History of receiving systemic chemotherapy or CAR-T therapy for ALL.

Impaired cardiac function, including any one of the following:

.LVEF <45% as determined by MUGA scan or echocardiogram. .Complete left bundle branch block. .Use of a cardiac pacemaker.

* ST depression of >1mm in 2 or more leads and/or T wave inversions in 2 or more contiguous leads. .Congenital long QT syndrome. .History of or presence of significant ventricular or atrial arrhythmia. .Clinically significant resting bradycardia (<50 beats per minute). .QTc >450 msec on screening ECG (using the QTcF formula). .Right bundle branch block plus left anterior hemiblock, bifascicular block. .Myocardial infarction within 3 months prior to starting olverembatinib . .Angina pectoris.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of olverembatinib or chidamide (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). .History of or current autoimmune disease. .History of or current relevant CNS pathology. .Presence of CNS leukemia. .History of or current autoimmune disease. .History of other malignancies. .Presence active infection.
* Nursing women or women of childbearing potential not willing to use an effective form of contraception during participation in the study and at least 3 months thereafter or male patients not willing to ensure effective contraception during participation in the study and at least three months thereafter.
* Not eigiable for this study, decided by PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete Molecular Response (CMR) | at 3 months
  CMR was defined as the absence of a detectable BCR::ABL1 transcript with a sensitivity of 0.01%.

SECONDARY OUTCOMES:
Overall survival (OS) | at 3 and 5 years
  OS was measured from time of study entry to the time of death or last follow-up
Event-free survival (EFS) | at 3 and 5 years
  EFS was measured from complete remission to the time of relapse or death
Adverse Events | at 1, 3 and 5 years
Event-free survival (EFS) of IKZF1del subgroup | at 3 and 5 years
Overall survival (OS) of IKZF1del subgroup | at 3 and 5 years
Event-free survival (EFS) of IKZF1plus subgroup | at 3 and 5 years
Overall survival (OS) of IKZF1plus subgroup | at 3 and 5 years
Event-free survival (EFS) of IKZF1plus/CD20 subgroup | at 3 and 5 years
Overall survival (OS) of IKZF1plus/CD20 subgroup | at 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hongsheng Zhou, M.D., Ph.D, Principal Investigator — Department of Hematology Nanfang Hospital; Zhixiang Wang, M.D., Ph.D, Study Director — Department of Hematology Nanfang Hospital; Ting Zhang, M.D., Ph.D, Study Director — Department of Hematology Nanfang Hospital; Ren Lin, M.D., Ph.D, Study Director — Department of Hematology Nanfang Hospital; Congcong Wang, Study Director — Department of Hematology Nanfang Hospital; Jiali Yao, Study Director — Department of Hematology Nanfang Hospital; Qianwei Liu, Ph.D, Study Director — Department of Hematology Nanfang Hospital
Locations (1):
- Dept of Hematology, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Foa R, Bassan R, Vitale A, Elia L, Piciocchi A, Puzzolo MC, Canichella M, Viero P, Ferrara F, Lunghi M, Fabbiano F, Bonifacio M, Fracchiolla N, Di Bartolomeo P, Mancino A, De Propris MS, Vignetti M, Guarini A, Rambaldi A, Chiaretti S; GIMEMA Investigators. Dasatinib-Blinatumomab for Ph-Positive Acute Lymphoblastic Leukemia in Adults. N Engl J Med. 2020 Oct 22;383(17):1613-1623. doi: 10.1056/NEJMoa2016272. PMID 33085860
- [Background] Jabbour E, Short NJ, Jain N, Huang X, Montalban-Bravo G, Banerjee P, Rezvani K, Jiang X, Kim KH, Kanagal-Shamanna R, Khoury JD, Patel K, Kadia TM, Daver N, Chien K, Alvarado Y, Garcia-Manero G, Issa GC, Haddad FG, Kwari M, Thankachan J, Delumpa R, Macaron W, Garris R, Konopleva M, Ravandi F, Kantarjian H. Ponatinib and blinatumomab for Philadelphia chromosome-positive acute lymphoblastic leukaemia: a US, single-centre, single-arm, phase 2 trial. Lancet Haematol. 2023 Jan;10(1):e24-e34. doi: 10.1016/S2352-3026(22)00319-2. Epub 2022 Nov 16. PMID 36402146

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT06220487/Prot_SAP_ICF_000.pdf